CLINICAL TRIAL: NCT03420079
Title: A Phase I, Multi-center, Open-label, Single-arm, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Anti-tumor Activities of FCN-411 Monotherapy in Advanced Non-small Cell Lung Cancer
Brief Title: A Phase I Study of FCN-411 in Advanced Non-small Cell Lung Cancer Chinese Patients With EGFR Positive Mutation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FCN001
Record Dates: First submitted 2017-11-14; First posted 2018-02-05 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
Keywords: advanced NSCLC; EGFR-TKI refractory
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: In the dose escalation cohort of FCN-411, the dose will be escalated from 4 mg, 8 mg, 16 mg, 24 mg to 32 mg. The MTD will be expanded to ascertain the RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation cohort of FCN-411 (Experimental): * FCN-411 will be orally administrated at five sequential dose levels, which are 4 mg, 8 mg, 16 mg, 24 mg, and 32 mg.
  * Patients must be diagnosed with locally advanced or metastatic NSCLC who have progressed following prior therapy with an EGFR TKI agent (+/- additional chemotherapy regimens).
  * Participants will receive FCN-411 monotherapy once daily (QD) for sequential 21-day cycles.
  Interventions: Drug: FCN-411 Dose-escalation
- Dose expansion cohort of FCN-411 (Experimental): * FCN-411 will be orally administrated at MTD.
  * Patients must be diagnosed with locally advanced or metastatic NSCLC who have progressed following prior therapy with an EGFR TKI agent (+/- additional chemotherapy regimens).
  * Participants will receive FCN-411 monotherapy once daily (QD) for sequential 21-day cycles.
  Interventions: Drug: FCN-411 Dose-expansion

INTERVENTIONS:
Drug: FCN-411 Dose-escalation — * FCN-411 is a pan EGFR inhibitor, which has strong activity against wild type (WT), HER2, HER4 and EGFR sensitive mutations (including but not limited to T790M and L858R mutation).
  * FCN-411 shows significant antitumor activity in a dose-dependent manner in in vivo models of lung cancer, esophageal cancer and pharyngeal squamous cell carcinoma mediated by EGFR.
  Other Names: EGFR-TKI
  Arms: Dose escalation cohort of FCN-411
Drug: FCN-411 Dose-expansion — * FCN-411 is a pan EGFR inhibitor, which has strong activity against wild type (WT), HER2, HER4 and EGFR sensitive mutations (including but not limited to T790M and L858R mutation).
  * FCN-411 shows significant antitumor activity in a dose-dependent manner in in vivo models of lung cancer, esophageal cancer and pharyngeal squamous cell carcinoma mediated by EGFR.
  Other Names: EGFR-TKI
  Arms: Dose expansion cohort of FCN-411

SUMMARY:
This phase I trial with dose-escalation stage and dose-expansion stage is the first-in-human study of FCN-411, a drug being developed for treatment of advanced cancers. The initial purpose of the study is to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of FCN-411 monotherapy in EGFR-positive mutation non-small cell lung cancer chinese patients. The study will also provide early information on how the body handles the drug (pharmacokinetics) and on the anti-tumor activities of FCN-411.

DETAILED DESCRIPTION:
This is a multicenter, open, single arm phase I clinical trial to explore the dose of FCN-411 in advanced lung cancer patients with disease progression after standard treatment or unsuitable for standard treatment and to expand the dose in advanced NSCLC patients who failed EGFR-TKI treatment. During the screening period, patients need to provide tumor tissue/ blood samples collected after their disease progression for tumor biomarker detection. In this study, the safety, tolerance and pharmacokinetic characteristics of FCN-411 were observed by dose escalation study and dose expansion study, and the antitumor activity of FCN-411 was preliminarily evaluated to determine maximal tolerated dose (MTD) and recommended phase 2 dose (RP2D). The phase I dose escalation study includes two stages: single dose stage and continuous dose stage; phase I dose expansion study is continuous dose administration.

The research cycle is made up of screening period (day-28-day-1), single administration period (7 days), continuous administration period (every 21 days, evaluated every 6 weeks, until disease progression, intolerable toxicity, death, decision of the investigator or voluntary withdrawal of the patient), end of treatment, EOT) visit, safety follow-up (30 days after the last administration), survival follow-up (survival follow-up every 3 months from the safety follow-up until the end of the study). The end of study is one year after the first administration of the last enrolled patient or the end of treatment (whichever is earlier).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older.
2. Histological or cytological confirmed diagnosed advanced or metastatic NSCLC.
3. Documentation of disease progression while on previous continuous treatment with first-line EGFR TKI; patients must have confirmation of tumor EGFR activating mutations (exon 19 del, or exon 21 ins) and T790M status by biopsy sample or optical microscopy.
4. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG).
5. Have a life expectancy of at least 12 weeks.
6. Have measurable disease based on RECIST v1.1. Note: previously irradiated not chosen, unless disease progression after irradiation.
7. Adequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   1. Neutrophils (absolute value) ≥ 1.5×10^9/L;
   2. Hemoglobin ≥ 90 g/L;
   3. Platelet ≥ 90×10^9/L;
   4. Serum total bilirubin ≤ 1.5× ULN（for Patients with Gilbert Syndrome, total bilirubin ≤ 3×ULN and bilirubin ≤ 1.5×ULN should be permitted）
   5. Aspartate aminotransferase、alanine aminotransferase ≤ 2.5×ULN; for patients with hepatic metastases, AST、ALT ≤ 5×ULN;
   6. Creatinine < 1.5×ULN creatinine clearance rate≥ 45 mL/min (Cockcroft Gault for calculating)
8. Female subjects have a negative urine or serum pregnancy.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Treatment with an EGFR TKI within 14 days or about 5 half-lives, whichever is the longer, of the first dose of study drug;
   2. Any cytotoxic chemotherapy, investigational agents or anticancer drugs for the treatment from a previous treatment regimen within 14 days of the first dose of study treatment;
   3. Major surgery within 4 weeks of the first dose of study treatment;
   4. Systemic irradiation including whole brain irradiation;
   5. Previously treated by EGFR-TKI for T790M (for example Osimertinib).
2. P-glycoprotein inducers (for example Rifampicin) or inhibitors (for example ritonavir) are required during the study.
3. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
4. Meningeal metastases or CNS metastasis received intervention or malignancy related epilepsy; brain metastases without symptom are eligible.
5. Any serious or uncontrolled systemic disease, including but not limited to:

   1. Uncontrolled hypertension;
   2. Active hemorrhage;
   3. Active infections including hepatitis B, or hepatitis C;
   4. Human immunodeficiency virus positive;
   5. Child Pugh C;
   6. Bullous or exfoliative skin diseases;
   7. Severe malnutrition;
   8. History of keratitis or ulcerative keratitis or dry eye;
   9. Uncontrolled large amount of third interstitial fluid retention;
   10. Other serious diseases or mental disorders or laboratory abnormalities.
6. Cardiac function and disease are consistent with the following:

   1. QTc> 470 milliseconds from 3 electrocardiograms (ECGs);
   2. Any clinically important abnormalities in rhythm;
   3. Any factors that increase the risk of QTc prolongation;
   4. Congestive heart failure ≥ grade 3 by New York Heart Association (NYHA);
7. Previous history with interstitial lung disease、drug-induced interstitial lung disease or radiation pneumonitis require hormone therapy, or other active interstitial lung diseases required treatments.
8. Lung function met one of the following criteria:

   1. Oxygen saturation ≤ 88%;
   2. The first second forced expiratory volume< 50% of the predicted value;
   3. Diffusion capacity for CO < 50% of the predicted value.
9. Dysphagia, or active digestive system diseases or medical conditions potentially affect FCN-411 absorption.
10. Hypersensitivity to FCN-411 or similar compounds or excipients.
11. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Cmax of FCN-411 following single dose. | PK blood samples are collected at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 120 hours post-dose.
  Cmax of FCN-411 following single dose.
AUC of FCN-411 following single dose. | PK blood samples are collected at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 120 hours post-dose.
  AUC of FCN-411 After Single Dosing.
Cmax of FCN-411 following multiple dosing. | The datas should be evaluated multiple times on the eighth day、fifteenth day of Cycle 1, first day、second day of Cycle 2. Each cycle is 21 days.
  Cmax of FCN-411 After multiple dosing.
AUC of FCN-411 following multiple dosing. | The datas should be evaluated multiple times on the eighth day、fifteenth day of Cycle 1, first day、second day of Cycle 2. Each cycle is 21 days.
  AUC of FCN-411 After Multiple Dosing.
Tmax of FCN-411 following single dose. | PK blood samples are collected at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 120 hours post-dose.
  Tmax of FCN-411 following single dose.
Tmax of FCN-411 following multiple dosing. | The datas should be evaluated multiple times on the eighth day、fifteenth day of Cycle 1, first day、second day of Cycle 2. Each cycle is 21 days.
  Tmax of FCN-411 following multiple dosing.
t1/2 of FCN-411 following single dose. | PK blood samples are collected at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 120 hours post-dose.
  t1/2 of FCN-411 following single dose.
t1/2 of FCN-411 following multiple dosing | The datas should be evaluated multiple times on the eighth day、fifteenth day of Cycle 1, first day、second day of Cycle 2. Each cycle is 21 days.
  t1/2 of FCN-411 following multiple dosing

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital chinese academy fo medical scienced, Beijing, China

REFERENCES:
- [Result] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Result] Wu YL, Zhou C, Hu CP, Feng J, Lu S, Huang Y, Li W, Hou M, Shi JH, Lee KY, Xu CR, Massey D, Kim M, Shi Y, Geater SL. Afatinib versus cisplatin plus gemcitabine for first-line treatment of Asian patients with advanced non-small-cell lung cancer harbouring EGFR mutations (LUX-Lung 6): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Feb;15(2):213-22. doi: 10.1016/S1470-2045(13)70604-1. Epub 2014 Jan 15. PMID 24439929
- [Result] Yang JC, Shih JY, Su WC, Hsia TC, Tsai CM, Ou SH, Yu CJ, Chang GC, Ho CL, Sequist LV, Dudek AZ, Shahidi M, Cong XJ, Lorence RM, Yang PC, Miller VA. Afatinib for patients with lung adenocarcinoma and epidermal growth factor receptor mutations (LUX-Lung 2): a phase 2 trial. Lancet Oncol. 2012 May;13(5):539-48. doi: 10.1016/S1470-2045(12)70086-4. Epub 2012 Mar 26. PMID 22452895
- [Result] Soria JC, Felip E, Cobo M, Lu S, Syrigos K, Lee KH, Goker E, Georgoulias V, Li W, Isla D, Guclu SZ, Morabito A, Min YJ, Ardizzoni A, Gadgeel SM, Wang B, Chand VK, Goss GD; LUX-Lung 8 Investigators. Afatinib versus erlotinib as second-line treatment of patients with advanced squamous cell carcinoma of the lung (LUX-Lung 8): an open-label randomised controlled phase 3 trial. Lancet Oncol. 2015 Aug;16(8):897-907. doi: 10.1016/S1470-2045(15)00006-6. Epub 2015 Jul 5. PMID 26156651
- [Result] Miller VA, Hirsh V, Cadranel J, Chen YM, Park K, Kim SW, Zhou C, Su WC, Wang M, Sun Y, Heo DS, Crino L, Tan EH, Chao TY, Shahidi M, Cong XJ, Lorence RM, Yang JC. Afatinib versus placebo for patients with advanced, metastatic non-small-cell lung cancer after failure of erlotinib, gefitinib, or both, and one or two lines of chemotherapy (LUX-Lung 1): a phase 2b/3 randomised trial. Lancet Oncol. 2012 May;13(5):528-38. doi: 10.1016/S1470-2045(12)70087-6. Epub 2012 Mar 26. PMID 22452896
- [Result] Katakami N, Atagi S, Goto K, Hida T, Horai T, Inoue A, Ichinose Y, Koboyashi K, Takeda K, Kiura K, Nishio K, Seki Y, Ebisawa R, Shahidi M, Yamamoto N. LUX-Lung 4: a phase II trial of afatinib in patients with advanced non-small-cell lung cancer who progressed during prior treatment with erlotinib, gefitinib, or both. J Clin Oncol. 2013 Sep 20;31(27):3335-41. doi: 10.1200/JCO.2012.45.0981. Epub 2013 Jul 1. PMID 23816963
- [Result] Wong AL, Sundar R, Wang TT, Ng TC, Zhang B, Tan SH, Soh TI, Pang AS, Tan CS, Ow SG, Wang L, Mogro J, Ho J, Jeyasekharan AD, Huang Y, Thng CH, Chan CW, Hartman M, Iau P, Buhari SA, Goh BC, Lee SC. Phase Ib/II randomized, open-label study of doxorubicin and cyclophosphamide with or without low-dose, short-course sunitinib in the pre-operative treatment of breast cancer. Oncotarget. 2016 Sep 27;7(39):64089-64099. doi: 10.18632/oncotarget.11596. PMID 27577069
- [Derived] Lin L, Pan H, Li X, Zhao C, Sun J, Hu X, Zhang Y, Wang M, Ren X, Luo X, Shan G, Hui AM, Wu Z, Liu H, Tian L, Shi Y. A phase I study of FCN-411, a pan-HER inhibitor, in EGFR-mutated advanced NSCLC after progression on EGFR tyrosine kinase inhibitors. Lung Cancer. 2022 Apr;166:98-106. doi: 10.1016/j.lungcan.2022.01.025. Epub 2022 Feb 3. PMID 35248866
- See also: ICH Topic E6 - Guideline for Good Clinical Practice: Consolidated guideline finalised (step 4) in May 1996. Adopted by CPMP, July 96, issued as CPMP/ICH/135/95/step 5, post step errata, July 2002. — https://www.ema.europa.eu/en/documents/scientific-guideline/ich-e6-r1-guideline-good-clinical-practice_en.pdf
- See also: ICH Topic E9 - Statistical Principles for Clinical Trials: Consensus guideline finalised (step 4) on 5th February1998. Adopted by CPMP, March 1998, issued as CPMP/ICH/363/96/step 5. — https://www.ema.europa.eu/en/documents/scientific-guideline/ich-e-9-statistical-principles-clinical-trials-step-5_en.pdf